CLINICAL TRIAL: NCT03239730
Title: Arterial pH Selectively Predicts ICU Transfer in Obese Patients With Acute Dyspnea Presenting to the Emergency Department: a Prospective Comparative Cohort Study
Brief Title: Arterial pH Selectively Predicts Intensive Care Unit Transfer From the Emergency Department in Obese Patients With Acute Dyspnea
Status: Completed | Type: Observational
Sponsor: Association pour la Formation du Personnel à la Medecine d'Urgence (Other)
Collaborators: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: pH acute dyspnea
Record Dates: First submitted 2017-08-01; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Dyspnea; Respiratory Failure
Keywords: dyspnea; pH; blood gas analysis; emergency department; Intensive care unit
MeSH Terms: conditions — Dyspnea; Respiratory Insufficiency; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the prognostic value of arterial blood gas analysis in a cohort of Emergency Department patients presenting with shortness of breath of any cause, comparing obese and non-obese patients.

DETAILED DESCRIPTION:
Factors associated with admission to intensive care unit (ICU) or ED mortality before transfer to the ICU are analyzed in obese (BMI ≥ 30kg.m-2) and non-obese patients subgroups.

ELIGIBILITY:
Inclusion Criteria:

* patients who presented with acute dyspnea in the ED
* patients who had an ABG analysis as part of the ED standard management

Exclusion Criteria:

* Patients with treatment limitation decisions made by the medical teams against ICU admission, including severe cognitive impairment or palliative care ,
* Patients with immediate transfer to ICU due to shock and hemodynamic instability at ED admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was derived from a cohort of adult patients admitted to the ED with acute dyspnea
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2014-05-30 (Actual)

PRIMARY OUTCOMES:
Composite of admission to the ICU or in ED mortality before ICU admission | up to 1 day (direct admission to ICU from ED)
  Admission to the ICU following ED management will be at the discretion of the attending ICU physician, and in agreement with current guidelines for ICU admission, according to standard management

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha SEBBANE, MD, PhD, Principal Investigator — Emergency Department, University Hospital, Montpellier
Locations (1):
- Montpellier University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No